CLINICAL TRIAL: NCT07369466
Title: Preoperative Hippocampal Glucose Metabolism Levels and the Risk of Postoperative Delirium in Older Patients With Type 2 Diabetes: A Prospective Cohort Study
Brief Title: Association of Preoperative Hippocampal Glucose Metabolism With Postoperative Delirium in Older Diabetic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Chief Physician, Chinese PLA General Hospital
Other Study IDs: PLAGH-PET-01
Record Dates: First submitted 2026-01-10; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Delirium; Type 2 Diabetes
Keywords: Postoperative delirium; Type 2 Diabetes Mellitus; Positron-Emission Tomography; Hippocampus; Glucose metabolism
MeSH Terms: conditions — Emergence Delirium; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older T2DM Hepatectomy Cohort

SUMMARY:
Objective: To investigate the association between preoperative hippocampal glucose metabolism levels and the risk of postoperative delirium (POD) in elderly patients with type 2 diabetes (T2DM), and to provide a prospective neuroimaging biomarker for identifying high-risk populations.

Methods: This prospective cohort study plans to enroll 154 elderly T2DM patients scheduled for liver tumor resection at the First Medical Center of Chinese PLA General Hospital. Baseline cognitive function will be assessed using the Mini-Mental State Examination (MMSE) one day before surgery. Hippocampal glucose metabolism will be quantitatively evaluated by measuring the mean standardized uptake value (SUVmean) of bilateral hippocampi using ¹⁸F-FDG PET/CT. POD will be assessed twice daily from postoperative days 1 to 7 using the 3-Minute Diagnostic Interview for CAM (3D-CAM). The correlation between preoperative hippocampal SUVmean and POD incidence will be analyzed using univariate and multivariate logistic regression models. The predictive performance will be evaluated by constructing receiver operating characteristic (ROC) curves. Furthermore, the relationship between a peripheral insulin resistance marker (the triglyceride-glucose index, TyG index) and hippocampal metabolism levels will be analyzed.

Significance: This study aims to determine whether impaired preoperative hippocampal metabolism serves as an independent risk factor for POD. The findings are expected to provide a prospective functional neuroimaging biomarker for the early warning of POD and offer a theoretical basis for developing precise prevention strategies targeting cerebral metabolic abnormalities. This will facilitate the application of neuroimaging techniques in the field of perioperative brain dysfunction monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes mellitus (T2DM).
2. Age ≥ 65 years.
3. Scheduled for elective liver tumor resection surgery with an expected operative duration > 2 hours.
4. Underwent whole-body ¹⁸F-FDG PET/CT scan within 1 month prior to surgery.

Exclusion Criteria:

1. Patient declines to participate.
2. Inability to cooperate with cognitive assessments or a preoperative Mini-Mental State Examination (MMSE) score < 23.
3. American Society of Anesthesiologists (ASA) physical status classification ≥ IV.
4. History of organic brain disorders, including stroke, traumatic brain injury, or intracranial tumors.
5. History of psychiatric disorders or current use of antipsychotic medications.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This prospective cohort study will enroll elderly patients (age ≥ 65 years) diagnosed with type 2 diabetes mellitus (T2DM) who are scheduled for elective liver tumor resection surgery with an expected duration of >2 hours at the First Medical Center of Chinese PLA General Hospital. All participants will undergo preoperative ¹⁸F-FDG PET/CT scanning and cognitive assessment, and will be prospectively followed for the occurrence of postoperative delirium.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Delirium (POD) | From surgery completion to postoperative day 7
  Assessed by the 3-Minute Diagnostic Interview for CAM (3D-CAM), administered twice daily.

SECONDARY OUTCOMES:
Triglyceride-glucose (TyG) index | Within 7 days before surgery (preoperative baseline)
  Calculated as Ln [fasting triglycerides (mg/dL) × fasting glucose (mg/dL) / 2].

OTHER OUTCOMES:
Incidence of Postoperative Adverse Events within 30 Days | From surgery completion to postoperative day 30
  Incidence of postoperative adverse events within 30 days, including but not limited to cardiovascular adverse events, ischemic stroke, pulmonary infection, acute kidney injury, and pain assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, Professor, Study Chair — The First Medical Center of Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: Undecided
A data sharing plan has not been fully formulated yet and will be finalized prior to the completion of the study.